CLINICAL TRIAL: NCT01703611
Title: Diabetes in India Nutrition Guidelines Study (DINGS)
Acronym: DINGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Nutrition and Dietetics (Other)
Collaborators: Indian Institute of Nutritional Sciences (Unknown); Abbott Healthcare Private Limited (in India) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Academy-India-1; IINS-ANDF/2011/01 (Other: India Clinical Trial Registry)
Record Dates: First submitted 2012-10-06; First posted 2012-10-10 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Nutrition; Medical Nutrition Therapy; Diabetes Mellitus; Nutrition outcomes; Evidence Based Guidelines
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MNT according to AND EBNPG for Type 2 DM (Experimental): Six or more Medical Nutrition Therapy visits(education and counseling on diet, self management, and lifestyle changes) provided over a 12 month period according to Academy of Nutrition and Dietetic Evidence Based Nutrition Practice Guidelines (EBPGN) (www.guidelines.gov)
  Interventions: Other: MNT according to AND EBNPG for Type 2 DM
- Usual Nutrition Care (Active Comparator): Visits for usual nutrition therapy (diet and lifestyle changes) provided by dietitians over a 12 month period.
  Interventions: Other: Usual Nutrition Care

INTERVENTIONS:
Other: MNT according to AND EBNPG for Type 2 DM — Six or more Medical Nutrition Therapy visits(education and counseling on diet, self management, and lifestyle changes) provided over a 12 month period according to Academy of Nutrition and Dietetic Evidence Based Nutrition Practice Guidelines (EBNPG)(www.guidelines.gov)
  Other Names: Nutrition Counseling; Nutrition Care; Nutrition Therapy; Evidence Based Nutrition Practice
  Arms: MNT according to AND EBNPG for Type 2 DM
Other: Usual Nutrition Care — Usual nutrition care in India
  Other Names: Nutrition Counselling; Nutrition Therapy
  Arms: Usual Nutrition Care

SUMMARY:
A clinical trial to compare the patient outcomes from usual nutrition therapy by dietitians in India to patient outcomes from guideline-based Medical Nutrition Therapy (MNT).

DETAILED DESCRIPTION:
A cluster randomized clinical trial to compare patient outcomes from two different nutrition interventions by dietitians in India for persons with Type 2 Diabetes Mellitus (usual care vs Medical Nutrition Therapy provided according to the Academy of Nutrition and Dietetics Evidence-Based Nutrition Practice Guidelines)

ELIGIBILITY:
Inclusion and exclusion criteria for participant selection is listed both for the dietitians and patient participants.

Dietitian Participant

Inclusion Criteria:

* RD and Indian ICC CDE RD
* Active practice (at least two years post-professional degree), with enough newly diagnosed type 2 DM patients or patients not seen by an RD for the previous year, to be able to recruit four to six of them into the study each week

  * Work in an Diabetes centers and hospital diabetes outpatient or private practice with diabetologist to provide medical oversight for study
  * Have written approval from immediate supervisor and diabetologist indicating that MNT visits can be provided without cost to research study in accordance with ADA EBNPG and data collection can be accommodated.
  * Have computer and internet access. Minimum requirements are Microsoft Internet Explorer 8.0 with 1024 x 768 screen resolution in 256 colors. The browser must be enabled for Java, JavaScript and cookies
  * Have stable internet connection (no prolonged periods without or frequent disruptions in internet service
  * Have land phone line and faxing capabilities
  * Able to provide data documentation electronically or in a paper format
  * Obtain approval from their facility's Independent Ethics Committee (equivalent to US Institutional Review Board) for participation in the study (if required by the institution)
  * Able to adjust the institution's habitual counseling session schedule and duration as required by the study protocol
  * Commit to attendance during the full course of face to face training for three days (including part of a weekend), to be held at Chennai, India, and participate in the Webinars and conference calls

Exclusion criteria:

* Small clientele of adult type 2 DM,
* Fewer than two years' active clinical practice experience post-professional degree,
* Unable to comply with the other inclusion criteria (see inclusion section above).

Patient Participant

Patients' Inclusion Criteria:

* Must be over 19 years of age
* Must have medical diagnosis for treatment of type 2 DM,
* Patient must agree to return for follow-up visits (or data collection visit) during the 12 months study period
* Not seen by RD for one year prior to being recruited to the study

Patients' Exclusion Criteria:

* Currently being seen by RD for MNT
* Participated in nutritional consults with RD in past year
* Having insulin prescribed for DM treatment at time of recruitment
* Pregnant or lactating at time of study
* History of end stage renal disease or renal insufficiency; history of CVA, CAD or MI; COPD; CHF; untreated depression; severe psychiatric illness; cancer diagnosis in previous two years or on-going radiation or chemotherapy treatment
* Unplanned surgery requiring more than one overnight stay in the hospital within the previous week to initial visit
* The presence of cognitive or physical limitations that preclude making lifestyle or dietary changes as assessed by the RD during the initial interview
* Unable to return to office for data collection at 6 and 12 months and unable to commit to follow-up visits for EBNPG.

Patient Dis-enrollment or Stop Point for Study Participation

Patient will no longer be in the study after he/she reports the onset of:

* End stage renal disease or renal insufficiency;
* CVA, CAD or MI;
* COPD;
* Depression, severe psychiatric illness;
* Cancer diagnosis and treatment;
* CHF;
* Unplanned surgery requiring more than one overnight stay in the hospital within the previous week;
* Pregnant,
* Any onset of cognitive or physical limitations that preclude making lifestyle or dietary changes per RD assessment during study period,
* Other acute/chronic complications that could exacerbate the patient's diabetic condition or general well-being.
* Physician starts injectable insulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HbAIc decrease | 6 months and 12 months

SECONDARY OUTCOMES:
Weight change | 6 month and 12 month

OTHER OUTCOMES:
Lipid panel | 6 month and 12 month
  Total Cholesterol, LDL Cholesterol, HDL Cholesterol and Triglycerides
Blood pressure | 6 months and 12 months
  Systolic and Diastolic change from baseline measure

CONTACTS AND LOCATIONS:
Overall Officials: Esther F Myers, PhD, Principal Investigator — Academy of Nutrition and Dietetics; Varsha (none), PhD, Principal Investigator — Shri Shradda Hospital; Naomi Trostler, PhD, Principal Investigator — Hebrew University
Locations (14):
- India (14):
  - Nagajuna Hospital, Vijayawada, Andhra Pradesh
  - Barman Diabetes Specialties, Guwahati, Assam
  - Dia Care 1 & 2, Ahmedabad, Gujarat
  - Fortis Escorts Hospital, Faridabad, Haryana
  - Asian Institute of Medical Sciences, Faridabad, Haryana
  - Malabar Institute of Medical Sciences, Calicut, Kerala
  - Caritis Hospital, Kottayam, Kerala
  - BhaktiVedanta Hospital, Mumbai, Maharashtra
  - Star Hospitals, Hyderabad, Pradesh
  - Santokba Durlabji Memorial Hospital, Jaipur, Rajasthan
  - Sundaram Medical Foundation, Chennai, Tamil Nadu
  - PSG Hospitals, Coimbatore, Tamil Nadu
  - Sanjay Gandhi Post Graduate Institute, Lucknow
  - Fortis Hospital, Uttar Pradesh